CLINICAL TRIAL: NCT06132971
Title: Multi-court Trial of NBP to Prevent Substance Abuse and Mental Health Disorders
Brief Title: Multi-court Trial of NBP to Prevent Substance Abuse and Mental Health Disorders (MTC)
Acronym: MTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Irwin Sandler, Principal Investigator, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01 DAO26874-01A1
Record Dates: First submitted 2018-07-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Divorce; Drug Abuse; Mental Health Disorder
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All data was collected by trained interviewers or teachers. All data collectors were masked as to study conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP2 (Active Comparator): Participants were assigned to the 2-session New Beginnings Program intervention
  Interventions: Behavioral: New Beginnings Program
- NBP10 (Experimental): Participants were assigned to the 10-session New Beginnings Program
  Interventions: Behavioral: New Beginnings Program

INTERVENTIONS:
Behavioral: New Beginnings Program

SUMMARY:
This application requests funding to conduct a randomized effectiveness trial of The New Beginnings Program (NBP) delivered through a partnership of domestic relations courts, community service providers and the NBP research team. This is the first attempt to offer the population of families seeking divorce an evidence-based prevention program shown to have long-term effects on youth problem outcomes. It is estimated that over a third of U.S. children experience parental divorce, which confers elevated risk for multiple problems in childhood and adulthood including substance use and abuse, smoking, mental health problems, high risk sexual behavior, and physical health problems. Efficacy trials of the NBP found positive effects at post-test, 6-year and 15-year follow-ups. For example, at 6-year follow-up the participation in NBP led to reductions in marijuana, drug and alcohol use and a 37% reduction in prevalence of diagnosed mental disorder; and reductions in externalizing problems, internalizing problems and high risk sexual behavior. Positive effects also occurred for grade point average (GPA) and self esteem. For many of the effects of the NBP, the effects were stronger for youth who were at higher risk at program entry. Many of the program effects were mediated through the program effects to strengthen parenting. Funded by an Advanced Center for Intervention and Services Research grant (NIMH P30 MH068685) the investigators modified the NBP to translate it from a prototype tested in efficacy trials into a program that can be effectively delivered by community service providers and one that is appropriate across diverse cultural groups, and fathers as well as mothers. Pilot testing of the modified NBP and training and monitoring systems has demonstrated that they are highly acceptable to parents and providers. The investigators also developed and experimentally tested a system of parent recruitment that was found to be effective in getting parents to enroll (sign up to participate) in the NBP but, similar to other prevention parenting programs, initiation (attendance at one or more sessions) in the NBP in the pilot was low.

DETAILED DESCRIPTION:
SPECIFIC AIMS This application requests funding to conduct a randomized effectiveness trial of The New Beginnings Program (NBP), a prevention program for divorced families, as delivered through a partnership of domestic relations courts, community service providers and the NBP research team. This partnership would be the first systematic attempt to offer the population of families seeking divorce an evidence-based prevention program shown to have long-term effects to reduce youth problem outcomes. It is estimated that over a third of U.S. children experience parental divorce which confers elevated risk for multiple problems in childhood, adolescence and adulthood including substance use and abuse, cigarette smoking, mental health problems, high risk sexual behavior, and physical health problems. When evaluated in efficacy trials, the NBP has been shown to have positive program effects at post-test, 6-year and 15-year follow-ups. For example, at 6-year follow-up the participation in NBP led to reductions in marijuana, drug and alcohol use; a 37% reduction in prevalence of diagnosed mental disorder; and reductions in externalizing problems, internalizing problems and high risk sexual behavior. Positive program effects also occurred for grade point average (GPA) and self esteem. For many of the short- and long-term effects of the NBP, the effects were stronger for youth who were at higher risk at program entry. Mediational analyses have shown that program effects on short-term and 6-year youth outcomes were mediated through the program effects to strengthen parenting. Funded by an Advanced Center for Intervention and Services Research grant (NIMH P30 MH068685) the investigators modified the NBP to translate it from a prototype tested in efficacy trials into a program that can be effectively delivered by community service providers and one that is appropriate for diverse cultural groups, a broad age range of youth, and fathers as well as mothers. The investigators also revised the methods for training, technical assistance and ongoing monitoring of implementation. Pilot testing of the modified NBP and training and monitoring systems has demonstrated that they are highly acceptable to parents and providers. The investigators also developed and experimentally tested a system of parent recruitment that builds on an infrastructure that exists in domestic relations courts in 46 states. This strategy was effective in getting parents to enroll (sign up to participate) in the NBP but, similar to other prevention parenting programs, initiation (attendance at one or more sessions) in the NBP in the pilot was low.

The Specific Aims are to:

1. Examine whether 1380 children in 920 divorcing families randomly assigned to the NBP or workshop controls, show greater improvement when assigned to the NBP on measures of positive parenting, youth substance use and mental health problems compared to controls. Assessments will occur at pre-test, post-test and 6-month follow-up. The study will also test whether program effects on youth outcomes at the 6-month follow-up are mediated by program-induced effects on positive parenting at post-test. This will be the first experimental evaluation of the effectiveness of an evidence-based parenting program to prevent substance use and mental health problems of youth from divorcing families when delivered through a partnership of the courts and community service providers.
2. Test whether the effects of the NBP are moderated by level of child risk at program entry, youth age, parent gender or parent's ethnicity [i.e., Mexican American (MA) vs. non-Hispanic Caucasians (NHW)]. Based on previous trials of the NBP, a significant program x baseline risk interaction is predicted with stronger program effects expected at higher levels of child risk. Because the program was modified and pilot tested to make it appropriate across ethnic groups, parent gender, and age of child, testing the interaction effect for these three variables is viewed as exploratory and no significant interactions are predicted.
3. Examine whether variability in implementation accounts for variability in parenting and youth outcomes. Multiple dimensions of implementation that have been found to relate to outcomes of prevention parenting programs will be measured (e.g., fidelity, group leader process quality, additive adaptation, participant responsiveness) and their unique contribution to program effects will be assessed. The investigators will also test whether gender or ethnicity moderate the relations between each dimension of implementation and outcomes.
4. Experimentally test whether a brief telephone engagement interview increases initiation (i.e. attending at least one session) relative to a standard informational contact. The effect of the engagement interview will be tested for the overall sample, and separately for males and females, and MA and NHW.

The results of this study have significant public health implications to reduce substance abuse and mental health problems of youth who experience parental divorce, a highly prevalent stressful event. Further, the proposed study addresses three issues that have substantial implications for the effectiveness of parent-focused preventive interventions: subgroup differences in program benefits, relations of dimensions of implementation to outcomes and engagement of parents in evidence-based parenting programs.

ELIGIBILITY:
Inclusion Criteria:

* Filing for divorce or modification of a divorce decree within the past two years
* If never married, being in court to establish or change a parenting time agreement following separation in the past two years
* Having at least one child aged 3 to 18 with whom the parent spends three or more hours each week or one overnight every other week
* Being able to complete the program and assessments in English
* Not being mandated to a parenting class by the Juvenile Court or Child Protective Services.

Exclusion Criteria:

* Parents who received a divorce more than two years prior and did not have any court involvement in the past two years.
* Parents who could not complete the program or assessments in English
* Parents were mandated to a parenting program by Child Protective Services of Juvenile Court

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2415 (Actual)
Dates: Start 2012-07-30 (Actual); Primary Completion 2015-08-04 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist Internalizing Problems | The time frame was the past month
  Parents completed the Child Behavior Checklist which has previously shown good reliability and validity (CBCL; Achenbach & Rescorla, 2001) for children aged 6 to 18 (α = .89 ) for internalizing, problems.
Brief Problem Monitor Internalizing | Time Frame was the past month
  Children aged 9 or older completed the Brief Problem Monitor (BPM; Achenbach, McConaughy, Ivanova, & Rescorla, 2011) to assess internalizing (six items, α = .79),
Child Behavior Checklist Externalizing Problems | The timeframe was the past month
  Parents completed the Child Behavior Checklist which has previously shown good reliability and validity (CBCL; Achenbach & Rescorla, 2001) for children aged 6 to 18 (α =.90, and .95 for externalizing problems)
Parent report of total child behavior problems | The time frame was the past month
  A single measure of parent total behavior problems was calculated as the sum of the T scores across parent report of total behavior problems from the CBCL and Pre-school CBCL across the broad age range (T. M. Achenbach, personal communication, 2015).
Brief Problem Monitor Externalizing | The time frame is past month
  Children aged 9 or older completed the Brief Problem Monitor (BPM; Achenbach, McConaughy, Ivanova, & Rescorla, 2011) to assess externalizing (seven items, α = .71).
Brief Problem Monitor Total Problems | The time frame is past month
  Children aged 9 or older completed the Brief Problem Monitor (BPM; Achenbach, McConaughy, Ivanova, & Rescorla, 2011) to assess total problems (19 items, α = .86).
Preschool Child Behavior Checklist Internalizing Problems | Past month
  Parents completed the Preschool Child Behavior Checklist (Pre-CBCL; Achenbach & Rescorla, 2000) for children aged 3 to 5 (α = .89) for internalizing problems)
Parent report of child internalizing problems | Past month
  T scores were calculated for CBCL and Pre-CBCL internalizing problem subscales based on child age and gender and combined to assess internalizing across the broad age range (T. M. Achenbach, personal communication, 2015).
Parent report of child externalizing problems | Past month
  Parents completed the Preschool Child Behavior Checklist (Pre-CBCL; Achenbach & Rescorla, 2000) for children aged 3 to 5 (α = .91 for externalizing problems).
Parent report of child externalizing problems | Past month
  Parent report of child externalizing problems was scored as the sum of T scores for the CBCL and Pre-CBCL externalizing subscales based on child age and gender and combined to assess internalizing, externalizing, and total problems across the broad age range (T. M. Achenbach, personal communication, 2015).

SECONDARY OUTCOMES:
Parent Report of Parent child relationship quality | Time frame was the past month
  Parent-child relationship quality was assessed using factor scores from a two-factor confirmatory factor analysis model. Indicators of parent-child relationship quality were involvement (six items, Menning, 2006), family routines (seven items, Jensen, et al., 1983), parent-child communication (10 items open communication subscale, Barnes and Olsen, 1982), closeness (single item, Stewart, 2003) and acceptance subscale of the CRPBI (16 items, Shaefer, 1965). The two-factor model closely fit the data at pretest, χ2 (17) = 69.8.
Parent Report of Rejection | Time frame was the past month
  We treated parent report of rejection as a separate measure because it did not load highly with the other indicators of parent-child relationship. Parent report of rejection was assessed using the rejection subscale of the CRPBI (16 items, Schaefer, 1965)
Monitoring | Time frame was the past month
  Parent report of monitoring as a separate measure because parents completed this measure only for children age 9 or older. Monitoring was assessed using the Child Monitoring Scale (11 items, Hetherington et al., 1992).
Parent report of Discipline | Time frame was the past month
  Parent report of discipline was assessed as a single measure which aggregated the scores from multiple indicators using factor scores from a two-factor confirmatory factor analysis model. The two-factor model closely fit the data at pretest, χ2 (17) = 69.8.
  Indicators of discipline that loaded on the discipline factor were consistency subscale of the CRPBI (16 items Schaefer, 1965), follow-through subscale of the Oregon Discipline Scale (11 items, Oregon Social Learning Center, 1991), and appropriate use of discipline (ratio) from the Oregon Discipline Scale (14 items. Oregon Social Learning Center).
Child report of positive parenting | Time Frame was the past month
  Child report of positive parenting was assessed as a single factor score which aggregated the scores from multiple indicators as the factor score based on a a confirmatory factor analysis which found that a single factor model had a good fit to the data χ2 (17) = 58.25, RMSEA = .07. CFI = .98. The indicators on this model were child reports of involvement (six items, Menning, 2006), family routines (7 items, Jensen et al., 1983), open communication subscale of the Parent-Adolescent Communication Scale (10 items, Barnes a\& Olson, 1982), closeness was measured using a single item (Stewart, 2003), the acceptance subscale of the CRPBI (16 items, Schaefer, 1965), the rejection subscale of the CRPBI (16 items, Schaefer, 1965), the consistency of discipline subscale of the CRPBI (8 items, Schaefer, 1965), and the Child Monitoring Scale (11 items, Hetherington et al., 1992).

OTHER OUTCOMES:
Parent report of Interparental conflict | Past month
  Parents reported on interparental conflict using four items from the Children's Perception of Interparental Conflict (α = ..90) ((Grych, Seid, & Fincham, 1992).
Child report of exposure to interparental conflict | Past month
  Children reported on exposure to interparental conflict using 13 items from the Children's Parent Interparental Conflict scale (Grych, Seid & Fincham, 1992) and two items developed for this study to assess parents arguing in from of them (α = ..87)
Child report of being caught in the middle | Past month
  Children report on being caught in the middle of their parents arguments using a nine item scale. Seven of the items on this scale were from the Caught in the Middle Scale (Buchanan, Maccoby & Dornbusch, 1991). Two items from this scale were child reports of their exposure to badmouthing from the Divorce Events Schedule Child (Sandler, Wolchik & Braver, 1988). Reliability of this single nine item scale was good ((α = ..78).

CONTACTS AND LOCATIONS:
Locations (1):
- Sharlene Wolchik, Tempe, Arizona, United States